CLINICAL TRIAL: NCT01489800
Title: The Impact of Early Feeding After Radical Cystectomy for Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAI0046
Record Dates: First submitted 2011-12-08; First posted 2011-12-12 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Bladder Cancer; Complications
Keywords: feeding; complications; radical cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Feeding (Experimental): Introduction of clear liquid diet 24 hours after extubation with advancement to regular diet 24 hours thereafter if there is no significant nausea or vomiting.
  Interventions: Behavioral: Clear liquid diet
- Control Feeding (No Intervention): Standard of care with introduction of clear liquid diet at time of return of bowel function as determined by flatus. Advancement to full diet 24 later if clear diet well tolerated.

INTERVENTIONS:
Behavioral: Clear liquid diet — clear liquid diet, the same for each arm, will be given 24 hours after extubation as the intervention in the experimental arm.
  Other Names: liquid diet
  Arms: Early Feeding

SUMMARY:
Complications after radical cystectomy for bladder cancer range from 30-40%, many of which are related to bowel function. Patients usually wait to eat until return of bowel function, although there is evidence that after primary intestinal or colonic surgery, patients may take food ad lib immediately, and that this is is associated with lower complication rate and shorter length of stay. The investigators hypothesize that early access to oral enteral nutrition (food at will) after cystectomy and urinary diversion will reduce the complication rate both in-hospital and within 90 days after hospital discharge.

DETAILED DESCRIPTION:
Subjects preparing to undergo radical cystectomy and urinary diversion for bladder cancer that provide informed consent will be randomized into 1 of 2 study arms. The experimental arm will be offered clear liquid diet 24 hours after extubation and advanced to regular diet 24 hours later if clear liquids are well tolerated. The standard/control arm will receive a clear liquid diet at the time of return of bowel function, determined by significant flatus or bowel movements.

Information related to time to return of bowel function, frequency of nausea/vomiting, hospital complications and length of stay will be recorded. Patients will be followed with phone calls and chart reviews at 30, 60 and 90 days following surgery. Additional hospital admissions and/or complications will be determined with those phone calls.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18
* Bladder cancer
* Elect radical cystectomy and urinary diversion as treatment
* Able to provide informed consent

Exclusion Criteria:

* Radical cystectomy for reason other than bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Complication rate | 90 day
  powered to detect 50% reduction in complication rate, from 40% down to 20%

SECONDARY OUTCOMES:
Primary Hospital Length of Stay | 30 days
  time from admission for surgery until discharge after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell C. Benson, M.D., Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - New York Hospital - Cornell, New York, New York
  - Columbia Univeristy Medical Center, New York, New York

REFERENCES:
- [Background] Chang SS, Cookson MS, Baumgartner RG, Wells N, Smith JA Jr. Analysis of early complications after radical cystectomy: results of a collaborative care pathway. J Urol. 2002 May;167(5):2012-6. PMID 11956429
- [Background] Lassen K, Kjaeve J, Fetveit T, Trano G, Sigurdsson HK, Horn A, Revhaug A. Allowing normal food at will after major upper gastrointestinal surgery does not increase morbidity: a randomized multicenter trial. Ann Surg. 2008 May;247(5):721-9. doi: 10.1097/SLA.0b013e31815cca68. PMID 18438106
- [Background] Pruthi RS, Nielsen M, Smith A, Nix J, Schultz H, Wallen EM. Fast track program in patients undergoing radical cystectomy: results in 362 consecutive patients. J Am Coll Surg. 2010 Jan;210(1):93-9. doi: 10.1016/j.jamcollsurg.2009.09.026. Epub 2009 Oct 28. PMID 20123338
- [Result] Deibert CM, Silva MV, RoyChoudhury A, McKiernan JM, Scherr DS, Seres D, Benson MC. A Prospective Randomized Trial of the Effects of Early Enteral Feeding After Radical Cystectomy. Urology. 2016 Oct;96:69-73. doi: 10.1016/j.urology.2016.06.045. Epub 2016 Jul 8. PMID 27402372